CLINICAL TRIAL: NCT03762928
Title: A PHASE 1, RANDOMIZED, OPEN LABEL, 2-WAY CROSSOVER STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSE PF-06651600 ON THE PHARMACOKINETICS OF SINGLE DOSE MIDAZOLAM AND EFAVIRENZ IN HEALTHY PARTICIPANTS
Brief Title: ESTIMATION OF THE EFFECT OF MULTIPLE DOSE PF-06651600 ON THE PHARMACOKINETICS OF SINGLE DOSE MIDAZOLAM AND EFAVIRENZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7981017
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects
Keywords: PK; Phase 1
MeSH Terms: interventions — PF-06651600; Midazolam; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- midazolam/efavirenz (Experimental)
  Interventions: Drug: midazolam; Drug: efavirenz
- PF-06651600/midazolam/efavirenz (Experimental)
  Interventions: Drug: PF-06651600; Drug: midazolam; Drug: efavirenz

INTERVENTIONS:
Drug: PF-06651600 — 200 milligram (mg) PF-06651600 once daily (QD) orally for 11 days
  Arms: PF-06651600/midazolam/efavirenz
Drug: midazolam — single administration of midazolam 2 mg oral solution
Drug: efavirenz — single administration of efavirenz 50 mg capsule

SUMMARY:
The current study will estimate any inhibitive or inductive effect of PF-06651600 on the pharmacokinetics of midazolam and efavirenz.

ELIGIBILITY:
Inclusion Criteria:

Male and female participants who are healthy Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease
* Any condition possibly affecting drug absorption
* Known immunodeficiency.
* Infection with hepatitis B or hepatitis C viruses
* acute or chronic infections or infection history judged to be clinically significant by the investigator
* History of any lymphoproliferative disorder
* known present or a history of malignancy other than a successfully treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* live (attenuated) vaccines within 6 weeks prior to the first dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-01-27 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
single dose Area under the curve at last quantifiable infinity time of midazolam | Hour 0, 0,5, 1, 2, 4, 6, 8, 12, 16, 24 hours post-dose
Single dose Area under the Curve from time 0 to 72 hours post-dose of efavirenz | hour 0, 0,5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose

SECONDARY OUTCOMES:
number of subjects with significant change from baseline in vital signs | hour 0 on study days 1, 4, 10 and 13 post-dose
number of subjects with significant change from baseline in laboratory safety tests results | study days -1, 4, 13 post-dose
number of subjects with treatment emergent adverse events (TEAE) | Baseline up to 35 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981017&StudyName=A+Phase+1%2C+Randomized%2C+Open+Label%2C+2-way+Crossover+Study+To+Estimate+The+Effect+Of+Multiple+Dose+Pf-06651600+On+The+Pharmacokinetics+Of+Single+Dose+Midazolam+And+Efavirenz+In+Healthy+Participants